CLINICAL TRIAL: NCT06097312
Title: Prospective, Observational, Non-interventional Study Designed to Detect and Describe Pregnancy Outcomes in Women Exposed to PREHEVBRIO® [Pregnancy Outcomes Registry]
Brief Title: PREHEVBRIO Pregnancy Outcomes Registry
Status: Recruiting | Type: Observational
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PREHEVBRIO-REGISTRY-US
Record Dates: First submitted 2023-09-28; First posted 2023-10-24 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Vaccine Exposure During Pregnancy
Keywords: PREHEVBRIO; Hepatitis B vaccine; Pregnancy
MeSH Terms: conditions — Hepatitis B | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Pregnant women who received PREHEVBRIO® vaccine within 28 days prior to conception or at any time during pregnancy.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The schedule of office visits and all treatment regimens will be determined by the treating health care provider. No interventions are administered as part of this protocol (observational study).

SUMMARY:
The registry is an observational surveillance program designed to recruit and encourage participation of women who were exposed to PREHEVBRIO® hepatitis B vaccine during pregnancy and to collect and analyze information related to post-exposure pregnancy and fetal and neonatal outcomes.

The objective of the Registry is to monitor and evaluate all received reports of PREHEVBRIO® vaccine exposure within 28 days prior to conception or at any time during pregnancy and delivery, as well as maternal, obstetrical, pregnancy, fetal and neonatal outcomes. This registry is primarily descriptive and designed to detect potential safety signals rather than test hypotheses.

DETAILED DESCRIPTION:
VBI Vaccines was granted a Biologic License by the FDA on 30 November 2021, to introduce PREHEVBRIO® in the United States for prevention of infection caused by all known subtypes of hepatitis B virus in adults 18 years of age and older. The vaccine has also been approved in the United Kingdom, Europe, Canada, and Israel, and is currently marketed in the United States, United Kingdom, the Netherlands, Belgium, and Israel.

According to the American College of Obstetricians and Gynecologists, pregnant women who are negative for hepatitis B virus infection and who are at risk for hepatitis B virus infection should be specifically targeted for hepatitis B vaccination. However, more data is required to make such a recommendation for PREHEVBRIO®. The rationale to conduct this study, include: (1) PREHEVBRIO®, as a newly licensed vaccine in the U.S., is not indicated for pregnant women; (2) pregnant women were actively excluded from trials during clinical development of PREHEVBRIO®; and (3) there have only been limited human data to inform the safety of PREHEVBRIO® administered during pregnancy. Since PREHEVBRIO® vaccination is not indicated in pregnancy, exposure to PREHEVBRIO® in pregnancy is likely to be inadvertent and to occur in early pregnancy.

The purpose of the registry is to detect, describe, and evaluate adverse pregnancy outcomes in females exposed to PREHEVBRIO® within 28 days prior to conception or at any time during pregnancy and to detect adverse fetal and/or neonatal outcomes at delivery or early termination.

The registry is strictly observational; schedule of office visits and all treatment regimens will be determined by the treating health care provider; no additional laboratory tests or assessments are required as part of this registry; only data noted as part of routine care will be collected. Subjects will be followed from enrollment until 3 months post-delivery or early termination of pregnancy.

Pregnant women will be enrolled in the registry prospectively (after exposure to the product but before the conduct of any prenatal tests that could provide knowledge of the outcome of pregnancy). If the condition of the fetus has already been assessed through prenatal testing (e.g., targeted ultrasound, amniocentesis, etc.), such reports will be considered retrospective reports. Retrospective reports are also eligible for the registry, but they will be analyzed separately from prospective reports. The analyses of study data will primarily use descriptive and inferential statistical methods designed to detect potential safety signals, rather than test hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman who received PREHEVBRIO® vaccine within 28 days prior to conception or at any time during pregnancy. The time of conception will be calculated as the most reliable estimated date of delivery (EDD) minus 38 weeks. For this registry, gestational weeks will be estimated from the EDD or as corrected EDD, if a more reliable EDD (e.g., by ultrasound) is provided. If the EDD is not available or never estimated, the first day of the last menstrual period (LMP) will be used to estimate gestational age and EDD.
* The subject provided consent prior to enrollment (for eligible subjects under 18 years old, consent must be obtained from the subject's legally authorized representative).
* The subject documents agreement with the release of medical information and contact with her healthcare providers (e.g., PCP, obstetrician, nurse midwife) and the infant's healthcare provider (e.g., pediatrician) for the purpose of collecting medical information.
* Reporter's (participant and/or healthcare provider) contact information is available to allow for follow up.

Exclusion Criteria:

* Subjects participating in another investigational device or drug study product within 28 days prior to conception or at any time during pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who received PREHEVBRIO® vaccine within 28 days prior to conception or at any time during pregnancy are eligible for inclusion. Because the vaccine is not indicated in pregnancy, the majority of exposures are likely to be inadvertently administered during the first trimester of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of spontaneous abortion | Less than 20 weeks of gestation, measured from the day of conception to the day of abortion
  Pregnancy loss <20 weeks of gestation
Rate of major congenital malformations | From enrollment until 3 months post-delivery
  Major structural or genetic birth defects, including conditions that (1) result from a malformation, deformation, or disruption in one or more parts of the body, a chromosomal abnormality, or a known clinical syndrome; (2) are present at birth; and (3) have a serious, adverse effect on health, development, or functional ability

SECONDARY OUTCOMES:
Rate of pre-term birth | From enrollment until delivery
  Infant born at gestational age <37 weeks of gestation
Rate of term labor | From enrollment until delivery
  Infant born at gestational age ≥37 weeks of gestation
Rate of fetal death/stillbirth | 20 or more weeks of gestation, measured from the day of conception to the day of fetal death/stillbirth, up to 10 months
  Pregnancy loss ≥20 weeks of gestation
Rate of induced abortion | From gestation until termination of pregnancy, up to 10 months
  Voluntary interruption of pregnancy, including pregnancy termination that occurs electively, to preserve maternal health, or due to fetal abnormalities
Rate of ectopic pregnancy | From gestation until termination of pregnancy, up to 10 months
  An ectopic pregnancy occurs when a fertilized egg grows outside of the uterus
Rate of low birth weight | From enrollment until delivery
  Infant born with birth weight <2500 g
Rate of major congenital abnormalities | From enrollment until 3 months post-delivery
  Includes transient defects, chromosomal abnormalities, genetic syndromes, and/or positional defects that are prematurity related

CONTACTS AND LOCATIONS:
Locations (1):
- ProPharma, Recruiting Nationwide, Overland Park, Kansas, United States